CLINICAL TRIAL: NCT06069154
Title: Percutaneous Cryoneurolysis: A Single-administration, Non-opioid, Non-addictive, Multiple-month Analgesic for Thoracic Trauma Free of Systemic Side Effects
Brief Title: Ultrasound-Guided Percutaneous Cryoneurolysis to Treat Pain Following Thoracic Trauma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRYO for Trauma (DoD)
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Rib Fracture; Rib Fracture Multiple
MeSH Terms: conditions — Rib Fractures | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicenter, randomized, triple-masked, sham-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individual who performs the procedure (and will not have subsequent contact with the participant).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis (Active Comparator): Active cryoneurolysis of the intercostal nerve of each fractured rib along with one cephalad and one caudad will be targeted: for each nerve the cryoneurolysis device will be triggered using 3 cycles of 2-minute nitrous oxide activation separated by 1-minute defrost periods (Epimed) or for the Varian: 5.5-minute [all but 5 participants] or 3-minute [5th - 12th participants; changes based on new laboratory and subsequently clinical data] argon activation (2000 psi starting at 100% power but decreased to keep return gas flow temperature warmer than -100C) followed by a 30-second helium defrost. For the active comparator, the gas will be deployed to the tip where a drop in temperature will result in cryoneurolysis.
  Interventions: Device: Cryoneurolysis; Procedure: Sham peripheral nerve block
- Sham Procedure (Sham Comparator): Sham cryoneurolysis of the intercostal nerve of each fractured rib along with one cephalad and one caudad will be targeted: for each nerve the cryoneurolysis device will be triggered using 3 cycles of 2-minute nitrous oxide activation separated by 1-minute defrost periods (Epimed) or for the Varian: 1 cycle of 5.5 minutes [all but 5 participants] or 3 minutes [5th - 12th participants; changes based on new laboratory and subsequently clinical data] of argon and 30 seconds of helium. However, for the sham comparator, the gas will NOT be deployed to the tip, there there will NOT be a drop in temperature, and NO cryoneurolysis will occur.
  Interventions: Procedure: Local anesthetic peripheral nerve block; Device: Sham Cryoneurolysis

INTERVENTIONS:
Device: Cryoneurolysis — Active cryoneurolysis of the intercostal nerve of each fractured rib along with one cephalad and one caudad will be targeted: for each nerve the cryoneurolysis device will be triggered using 3 cycles of 2-minute nitrous oxide activation separated by 1-minute defrost periods (Epimed) or for the Varian: 5.5-minute [all but 5 participants] or 3-minute [5th - 12th participants; changes based on new laboratory and subsequently clinical data] argon activation (2000 psi starting at 100% power but decreased to keep return gas flow temperature warmer than -100C) followed by a 30-second helium defrost. For the active comparator, the gas will be deployed to the tip where a drop in temperature will result in cryoneurolysis.
  Other Names: cryoablation
  Arms: Cryoneurolysis
Procedure: Local anesthetic peripheral nerve block — Due to the pragmatic design of this trial, study participation will not alter an institution's current practice. Examples of peripheral nerve blocks include paravertebral, erector spinae plane, and serratus anterior nerve blocks. The injectate through the introducer will depend on the treatment group: for participants of the control group, ropivacaine 0.5% or bupivacaine 0.375% (both with epinephrine 1:400,000) will be injected (volume determined by institutional standard-of-care). This will provide a peripheral nerve block for the control group.
  Arms: Sham Procedure
Device: Sham Cryoneurolysis — Sham cryoneurolysis of the intercostal nerve of each fractured rib along with one cephalad and one caudad will be targeted: for each nerve the cryoneurolysis device will be triggered using 3 cycles of 2-minute nitrous oxide activation separated by 1-minute defrost periods (Epimed) or for the Varian: 1 cycle of 5.5 minutes [all but 5 participants] or 3 minutes [5th - 12th participants; changes based on new laboratory and subsequently clinical data] of argon and 30 seconds of helium. However, for the sham comparator, the gas will NOT be deployed to the tip, there will NOT be a drop in temperature, and NO cryoneurolysis will occur.
  Other Names: sham cryoablation
  Arms: Sham Procedure
Procedure: Sham peripheral nerve block — Due to the pragmatic design of this trial, study participation will not alter an institution's current practice. Examples of peripheral nerve blocks include paravertebral, erector spinae plane, and serratus anterior nerve blocks: for participants allocated to the cryoneurolysis group (experimental group), normal saline will be injected for the peripheral nerve block. This will result in a sham/placebo nerve block for the experimental group.
  Arms: Cryoneurolysis

SUMMARY:
Thoracic trauma frequently involve rib fractures which can be very painful for 2-3 months. Unfortunately, pain is not simply a "symptom" of the injuries, but a significant cause of additional medical problems: pain causes people to breath and cough less deeply/often which increases the risk of collapsing little parts of the lung. These collapsed areas often lead to complications which can increase the risk of death. In addition, the higher the amount of pain in the weeks following the fracture, the higher the risk of developing persistent, chronic pain that can last indefinitely. So, providing excellent pain control is very important for a variety of reasons. Various nerve blocks can greatly decrease pain, but even the longest acting are measured in hours or days, and not the weeks and months for which rib fracture pain can last. Therefore, opioids-"narcotics"-are the most common pain control method provided to patients; but they frequently do not provide enough pain control, have undesirable side effects like nausea and vomiting, and are sometimes misused which can lead to addiction or overdose.

A prolonged nerve block lasting multiple months from a single treatment may be provided by freezing the nerve using a process called "cryoneurolysis". With cryoneurolysis and ultrasound machines, a very small "probe" may be placed through anesthetized skin and guided to the target nerve to allow freezing. The procedure takes about 5 minutes for each nerve, involves little discomfort, has no side effects, and cannot be misused or addictive. After 2-3 months, the nerve returns to normal functioning. The investigators have completed a small study suggesting that a single cryoneurolysis treatment provides potent short- and long-term pain relief following thoracic trauma with rib fractures. The ultimate objective of the proposed research is to determine if percutaneous cryoneurolysis is an effective non-opioid, single-application treatment for pain following traumatic rib fracture.

The current project is a pragmatic, multicenter, randomized, triple-masked (investigators, participants, statisticians), sham/placebo-controlled, parallel-arm, human-subjects, post-market clinical trial to determine if cryoneurolysis is an effective non-opioid treatment for pain following traumatic rib fractures.

DETAILED DESCRIPTION:
The investigators propose a pragmatic, multicenter, randomized, triple-masked (investigators, participants, statisticians), sham/placebo-controlled, parallel-arm, human-subjects clinical trial to determine if cryoneurolysis is an effective non-opioid treatment for pain following traumatic rib fractures. Participants will be recruited at 6 enrolling centers:

* Brigham and Women's Hospital, Boston, Massachusetts
* University of Texas, Houston, Houston, Texas
* Massachusetts General Hospital, Boston, Massachusetts
* University of California, San Diego, San Diego, California
* Walter Reed National Military Medical Center, Bethesda, Maryland

For individuals of childbearing potential, a sample of urine will be collected before any study interventions to confirm a non-pregnant state [this is standard for any trauma regardless of study participation]. Participants will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied (blood pressure cuff, pulse oximeter, 5-lead ECG), and oxygen administered via a facemask. Midazolam and fentanyl (IV) will be titrated for patient comfort as needed throughout the procedure, while ensuring that patients remain responsive to verbal cues.

Treatment group allocation (randomization). Participants will be allocated to one of two possible treatments groups:

1. Cryoneurolysis
2. Local anesthetic nerve block (Control)

Randomization will be stratified by enrolling institution and fracture laterality (unilateral vs. bilateral) in a 1:1 ratio, and in randomly chosen block sizes. Randomization lists will be created using Statistical Analysis Software computer-generated tables by the informatics division of the Department of Outcomes Research (Cleveland Clinic, Cleveland, OH). Treatment group assignment will be conveyed to the enrolling sites via the same secure web-based system (RedCap) used to collect study endpoints. The investigator administering the study intervention will access the treatment group assignment using the secure web-based system and attach the appropriate probe to the cryoneurolysis device. Therefore, all investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the investigator and coordinator who perform the procedure (and will not have subsequent contact with the participant). This protocol will enable a randomized, triple-masked (including statistician), sham/placebo-controlled trial. It is impossible to mask the individuals performing the cryoneurolysis procedure because the ice ball forming at the distal end of the probe-with active treatment-is clearly visible by ultrasound; and the lack of an ice ball for placebo participants is equally clear. It is essential to continuously visualize the probe and target nerve throughout the two freeze/thaw cycles to ensure the entire nerve diameter is adequately treated and remains relatively motionless. This cannot be achieved if the ultrasound is turned off during nitrous oxide administration to mask the provider; and the investigators prioritize patient safety over masking of the physician administering the intervention.

All participants will be positioned seated or prone (investigator preference), have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied (blood pressure cuff, pulse oximeter, 5-lead ECG), and oxygen administered via a facemask. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The treatment sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol.

Peripheral nerve block. Due to the pragmatic design of this trial, study participation will not alter an institution's current practice. Examples of peripheral nerve blocks include paravertebral, erector spinae plane, and serratus anterior nerve blocks using a long-acting local anesthetic (ropivacaine or bupivacaine, both with epinephrine). The injectate through the introducer will depend on the treatment group: for participants allocated to the cryoneurolysis group (experimental group), normal saline will be injected for the peripheral nerve block. For participants of the control group, ropivacaine 0.5% or bupivacaine 0.375% (both with epinephrine 1:400,000) will be injected (volume determined by institutional standard-of-care). This will provide a placebo nerve block for the experimental group and actual peripheral nerve block for the control group.

Cryoneurolysis procedure. The intercostal nerve of each fractured rib along with one cephalad and one caudad will be targeted. For example, if ribs 3-5 are fractured, then the ipsilateral nerves for thoracic levels 2-6 will receive treatment. Using a linear- or curved-array transducer, the intercostal nerve will be visualized using ultrasound just inferior to each treated rib immediately distal to the costotransverse joint. A skin wheal of local anesthetic will be raised immediately inferior to the transducer to anesthetize the skin.

There are multiple types of cryoneurolysis machines cleared by the US FDA, all of which work on the same principle of a gas being passed through a small annulus, resulting in a dramatic pressure drop and accompanying temperature drop due to the Joule-Thomson effect. This study will utilize two different consoles: the Epimed International (Farmers Branch, TX) and Varian Medical Systems (Palo Alto, CA) machines. Which machine is used is determined simply by the machine that each enrolling center has at its disposal.

Varian: This machine uses argon for the freeze cycle and helium to help decrease the thaw period duration. Sham probes are not available for this type of machine, and therefore an active probe will be used for all participants. For participants randomized to active treatment, the probe placed in the patient will be triggered and the argon (and helium) passed through the probe and then back into the machine, and finally vented out from the console. For participants randomized to sham treatment, the probe in the patient will simply not be activated; instead, a second probe that is not inserted in the patient will be triggered which will create the same visual and auditory cues as for the active participants retaining the masked feature. The investigator administering the study intervention will access the treatment group assignment using the secure web-based system and activate the correct probe depending on the treatment group assignment. Therefore, all investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the unmasked investigator and coordinator who perform the procedure (and will not have subsequent contact with the participant).

Epimed: This machine uses nitrous oxide for the freeze cycle with a passive thaw (no gas flow). Cryoneurolysis probes are available that either (1) pass nitrous oxide to the distal end inducing freezing temperatures; or (2) vent the nitrous oxide at the proximal end of the probe so that no gas reaches the distal end, resulting in no temperature change. The latter is a sham procedure since without the temperature change, no ice ball forms and therefore the target nerve is not affected. Importantly, these probes are indistinguishable in appearance and will be differentiated only by an identifying stamp on the underside of the connector which is not visible during use. The investigator administering the study intervention will access the treatment group assignment using the secure web-based system and attach the appropriate probe to the cryoneurolysis device. Therefore, all investigators, participants, and clinical staff will be masked to treatment group assignment, with the only exception being the unmasked investigator and coordinator who perform the procedure (and will not have subsequent contact with the participant).

These protocols will enable a randomized, triple-masked (including statistician), sham/placebo-controlled trial. For both types of machines, it is impossible to mask the individuals performing the cryoneurolysis procedure because the ice ball forming at the distal end of the probe-with active treatment-is clearly visible by ultrasound; and the lack of an ice ball for sham participants is equally clear. It is essential to continuously visualize the probe and target nerve throughout the freeze/thaw cycle(s) to ensure the entire nerve diameter is adequately treated and remains relatively motionless. This cannot be achieved if the ultrasound is turned off during nitrous oxide or argon administration in an attempt to mask the provider; and the investigators prioritize patient safety over masking of the physician administering the intervention.

The cryoneurolysis sites will already be cleansed with chlorhexidine gluconate and isopropyl alcohol. The intercostal nerve of each fractured rib along with one cephalad and one caudad will be targeted. For example, if ribs 3-5 are fractured, then the ipsilateral intercostal nerves 2-6 will receive treatment. The intercostal nerve will be visualized using ultrasound just inferior to each treated rib immediately distal to the costotransverse joint. A skin wheal of lidocaine will be raised inferior to the transducer to anesthetize the skin.

A portable cryoneurolysis console device (Varian Medical Systems or Epimed International) will be used with the appropriate probe (either active or sham).

Varian: The probe will be inserted adjacent to the intercostal nerve. The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute [all but 5 participants] or 3-minute [5th - 12th participants; changes based on new laboratory and subsequently clinical data] argon activation (2000 psi starting at 100% power but decreased to keep return gas flow temperature warmer than -100C) followed by a 30-second helium defrost. The Varian machine provides its own timer so that the gas cycle timing is precise to the second. The probe will be withdrawn, and this process repeated for each additional intercostal nerve to be treated. For bilateral fractures, the study intervention will be repeated on the contralateral side with the same probe.

Epimed: The probe will be inserted adjacent to the intercostal nerve. The cryoneurolysis device will be triggered using 2 cycles of 2-minute gas activation (active or sham) separated by a 1-minute defrost. An observer (usually the research coordinator) will time the cycles and indicate to the investigator when the 2- & 1-minute periods have concluded to ensure adequate treatment duration. The probe will be withdrawn, and this process repeated for each additional intercostal nerve to be treated. For bilateral fractures, the study intervention will be repeated on the contralateral side with the same probe.

Post-treatment course. Standard local supplemental analgesics will be used due to the pragmatic design of this trial. For analysis purposes, all opioids will be converted to oral oxycodone equivalents. Following a cryoneurolysis treatment, no action is required by patients. For example, in contrast to epidural infusions, there is no infusion pump to manage or anesthetic fluid to replenish. Patients will be provided with a hand-held incentive spirometer to keep at their bedside both while admitted and at home. Participants will be instructed in their use based on the American Association of Respiratory Care (AARC) clinical practice guideline, and then use the spirometer unsupervised at least hourly.

Following study completion, the results will be mailed electronically or by the United States Postal Service to all enrolled participants in written form using non-technical (e.g., "layperson") language.

Statistical Plan.

Primary Aim: To determine the effect of cryoneurolysis on opioid requirements and analgesia following traumatic rib fracture.

Hypothesis 1: Cumulative opioid consumption will be decreased in the first 2 months with cryoneurolysis compared with usual and customary analgesia.

Hypothesis 2: Fracture pain will be decreased within the first 2 months with cryoneurolysis compared with usual and customary analgesia (measured with a Numeric Rating Scale).

Primary Objective (Hypotheses 1 and 2). The investigators will estimate the treatment effect of cryoneurolysis on opioid consumption (Hypothesis 1) and average pain score (Hypothesis 2) using a joint hypothesis-testing framework. The investigators will conclude that cryoneurolysis is more effective compared to the standard of care if it is noninferior on both opioid consumption and pain score, and superior for at least one of the outcomes during the first 2 months after the intervention. No adjustment for multiple testing is needed for noninferiority testing since the investigators require noninferiority on both pain score and opioid consumption outcomes.

Noninferiority Testing. Hypothesis 1 (Opioid consumption). Cumulative opioid assumption is typically log-normally distributed. The investigators will therefore assess the treatment effect on the log-transformed cumulative opioid consumption at 2 months using a linear regression model. The investigators will test for NI of cryoneurolysis to standard of care using a 1-tailed test assuming alpha of 0.025 and NI delta of 1.2 for the ratio of geometric means (treatment/placebo). All opioids will be converted to oral oxycodone equivalents.

Hypothesis 2 (Average pain score). The investigators will test for noninferiority (NI) of cryoneurolysis to standard of care using 1-tailed tests and assuming a 1-tailed alpha of 0.025. The primary pain outcome will be the area under the curve (AUC) of patient "average" pain scores over the first 2 months (60 days; AUC-60). For this outcome the noninferiority (NI) delta will be a ratio of geometric means of 1.2 in the AUC-60. Since AUC-60 is expected to be skewed and also to have some proportion of zero values, the investigators will estimate the treatment effect a 2-sample t-test on the log-transformed (AUC-60 + 1).177 Noninferiority will be concluded if the upper 95% confidence interval of the ratio of geometric means is below the NI delta, with P-value reported using a 1-tailed NI test [specific formula included in the IRB submission but format not enabled in this registry].

Superiority Testing. If NI is found on both pain and opioid use, the investigators will test for superiority on each of cumulative opioid consumption and average pain AUC-60 using 1-tailed tests (using the primary analyses specified above) with overall 1-tailed alpha of 0.025. Since there are 2 tests for superiority the investigators will apply a Holm-Bonferroni correction and use a significance criterion of 0.025/2 for the smaller P-value and 0.025 for the larger. Similar tests will be conducted for the sensitivity analyses for pain score. Cryoneurolysis will be concluded more effective at pain management than standard care, and the joint null hypothesis rejected, if found superior on at least pain score or opioid consumption and at least noninferior on both.

Secondary pain outcomes in first 60 days. For each of average, current, least and worst pain score the investigators will conduct all of the analyses describe above for average pain score, as well as 1) assessing the treatment-by-time interaction in a linear mixed effects model using all measurements over time, and 2) estimating and reporting the treatment effect at each time point while controlling type I error across time points within each outcome variable using the Holm-Bonferroni procedure.

Sensitivity analyses for average pain score methodology. In addition to analyzing the AUC, the investigators will assess the treatment effect on patient "average" pain scores over time using a linear mixed effects model assuming an autoregressive correlation structure across scores for the same individual over time. Factors will be intervention, time (categorical) and baseline average pain score. The investigators will then test for noninferiority with a 1-tailed t-test in which the numerator is the estimated treatment effect minus the NI delta of 1 point and the denominator is the standard error of the estimated treatment effect. In another sensitivity analysis, the investigators will use a mixed effects proportional odds model with an autoregressive correlation structure to assess the treatment effect on pain score as an ordinal outcome.

Secondary Aims: To determine the effect of cryoneurolysis on physical and emotional functioning and chronic pain following traumatic rib fracture.

Hypothesis 3: The maximum voluntary inspiratory volume will be improved within the first 2 months with cryoneurolysis as compared with usual and customary analgesia (measured with an incentive spirometer).

Hypothesis 4: Physical and emotional functioning will be improved within the first 2 months with cryoneurolysis as compared with usual and customary analgesia (measured with the Interference Domain of the Brief Pain Inventory).

Hypothesis 5: The incidence and intensity of chronic pain will be decreased at 6 and 12 months with cryoneurolysis as compared with usual and customary analgesia (measured with a Numeric Rating Scale).

Hypothesis 6: The incidence of pulmonary complications will be decreased in the first year with cryoneurolysis as compared with usual and customary analgesia.

Hypothesis 3 (Maximum voluntary inspired volume). The effect of the intervention on patient area under the curve (AUC-60) of maximum voluntary inhaled volume will be assessed using either a 2-tailed t-test or Wilcoxon rank-sum test (with results presented as median difference (95% CI)), as appropriate. Secondarily the investigators will use a linear mixed effects model assuming an autoregressive correlation structure over the same time period, with fixed effects for treatment, time and baseline maximum voluntary inhaled volume. The investigators will further analyze the outcome over the entire first 12 months in a linear mixed effects model and also compare the treatment groups at each time point, controlling type I error as specified in the primary objective under "Secondary pain outcomes in first 60 days".

Hypothesis 4 (Physical and emotional functioning). Physical and emotional functioning of patients will be assessed using the interference domain of the Brief Pain Inventory (BPI), and the effect of the intervention will be assessed over the first 2 months as in Hypotheses 2 and 3 -- using patient AUC as primary analysis and a linear mixed model adjusting for baseline BPI-Interference domain score as secondary. The investigators will further analyze the outcome over the entire first 12 months in a linear mixed effects model and also compare the treatment groups at each time point, controlling type I error as specified in the primary objective under "Secondary pain outcomes in first 60 days".

Hypothesis 5 (Chronic pain). The effect of the intervention on the maximum/worst pain (ordinal scale) experienced by patients at each of 6 and 12 months will be assessed by separate Wilcoxon rank-sum tests at each time point, with treatment effect estimated as median difference (95% CI). In addition, a proportional odds logistic regression analysis adjusting for clinical site will be conducted for each time point. Second, the effect of the intervention on presence of any pain (binary - yes/no) at each of 6 and 12 months will be assessed using chi-square analyses and relative risk (95% CI), as well as Cochran-Mantel-Haenszel tests stratified by clinical site.

Hypothesis 6 (Pulmonary complications). Pulmonary complications will be a composite of hypoxia, pneumonia, acute respiratory distress syndrome, pulmonary embolus, aspiration, pneumothorax, and empyema measured during the first 12 months. The outcome will be the proportion of patients experiencing at least one of the distinct complications beginning after the intervention; the treatment effect will be analyzed using chi-square analyses and relative risk (95% CI), as well as Cochran-Mantel-Haenszel tests stratified by clinical site. The investigators will descriptively report the incidences and treatment effect on each individual component of the composite outcome, and where feasible, analyze the effect of the treatment effect on each component as a tertiary analysis (exploratory - no inference will be made).

Study-wide Type I error control. The investigators will use a parallel gatekeeping procedure to control the study-wide type I error at 0.05. For this procedure the investigators therefore have prioritized (a priori) the study outcomes into 7 ordered sets (below). Analysis will proceed in that order, and testing will proceed through each "gate" to the next set if and only if at least one outcome in the current set reaches significance. The significance level for each set will be 0.05 times a cumulative penalty for non-significant results in previous sets (i.e., a "rejection gain factor" equal to the cumulative product of the proportion of significant tests across the preceding sets). Within a set, a multiple comparison procedure (Holm-Bonferroni correction) will be used as needed to control the type I error at the appropriate level. Although the first set represents the 1-tailed joint hypothesis tests for noninferiority and superiority at alpha=0.025, without modifying the joint hypothesis test the investigators will use the corresponding 2-tailed alpha level of 0.05 for the gatekeeping, as all other sets involve 2-tailed tests. Some of the outcomes listed in the gatekeeping table are overall assessments over repeated measures. As detailed in statistical methods, treatment effects may also be assessed at individual time points. Such assessments will proceed according to the gatekeeping framework such that 1) type I error will be controlled across repeated measurements, and 2) inference will not be made on outcome variables that are excluded from formal testing/inference due to the gatekeeping results.

Parallel gatekeeping procedure Sets: Time frame... Required to pass to next set

1. H1/H2 - Joint hypothesis - opioids and pain Requires: NI both, Superiority on at least one: 2 months... Reject joint H0 (1 joint test)
2. H3 - Maximum voluntary inhaled volume H4 - BPI interference subscale: 2 months... Significance on either outcome
3. H5 - Chronic pain: (1) incidence and (2) worst pain: 6 months...Significance on either outcome
4. H6 - Pulmonary complications: 12 months... Significance on either outcome
5. H5 - Chronic pain: (1) incidence and (2) worst pain: 12 months... Not applicable

SAMPLE SIZE DETERMINATION

Sample Size Justification and Power Analyses. Sample size calculations and power analyses for the full study were informed by estimates from the pilot trial. The investigators plan on having at least 90% power for rejecting the joint hypothesis test for the primary aim.

Opioids. In the pilot study (N=10), the median [quartiles] of cumulative opioid consumption over 60 days were 85 [0, 126] in the control group and 0 [0, 9] in the treatment group. The ratio of geometric means [95% CI] was 0.09 [0.00, 9.61] indicating a 91% observed relative percent reduction in cumulative opioid consumption at 60 days. The investigators observed a coefficient of variation (CV) of 1.4. Noninferiority: Based on data from the investigators' enrollment centers, the investigators estimate that the overall ratio of polytrauma to non-polytrauma patients will be approximately 60:40. The investigators expect the effect on opioid consumption in the non-polytrauma cases to be much higher than for polytrauma patients. In the investigators' pilot study the investigators observed a ratio of geometric means of 0.1 (treatment/placebo) at 2 months. Assuming no true difference in opioid consumption for polytrauma patients (i.e., ratio of geometric means of 1), and assuming that the ratio of polytrauma to non-polytrauma cases would be 60:40, the weighted geometric mean ratio would be 0.4. Assuming a geometric mean ratio of 0.58, a NI delta of 1.2, 1-tailed alpha of 0.025 and CV of 1.4 the investigators would have 95.5% power to reject the null hypothesis. Superiority: A sample size of 60 patients in each group would yield 95.1% power to detect a geometric mean ratio of 0.46 (treatment/placebo), assuming a CV of 1.4, and 1-tailed alpha of 0.0125. The investigators will enroll up to 50 additional participants to allow for dropouts between enrollment and randomization. Therefore, a maximum total of 170 participants will be enrolled.

Pain. In the pilot study (N=10), the median [quartiles] of AUC pain scores from 2 to 60 days were 30 [4, 57] for cryoanalgesia and 263 [226, 336] for control, with difference in means (95% CI) of -262 (-413, -112) and ratio of geometric means (95% CI) of 0.06 (0.01, 0.41), indicating a 94% observed relative percent reduction in AUC pain through 60 days. The coefficient of variation (CV) for the log-transformed AUC was 1.23. Noninferiority: Assuming a true ratio of geometric means in AUC-60 of 0.62, a NI delta of 1.2, 1-tailed alpha of 0.025 and CV of 1.2, a sample size of 60 patients per group would yield 95.6% power to detect noninferiority. Superiority: A sample size of 60 patients in each group would yield 95.3% power to detect a geometric mean ratio of 0.52, assuming a CV of 1.2, and 1-tailed alpha of 0.0125. With the same sample size, the investigators would have 92% power to detect a decrease of 1.3 points in pain score in a linear mixed effects model (sensitivity analysis) assuming a mean difference of 0, 1-tailed alpha of 0.0125, intraclass correlation (ICC) of 0.63, standard deviation of 2.5, and an average cluster size (number of measurements per subject) of 10.

Power for Joint Hypothesis testing. The investigators will have 90% power to reject the joint null hypothesis; e.g, 95% power for superiority on pain times 96% power for NI on opioids = 91%, assuming independence.

Polytrauma cases (%) Polytrauma cases - geom. mean ratio (treatment/placebo) Non-polytrauma cases (%) Non-polytrauma cases - geom. mean ratio(treatment/placebo) Weighted geometric mean ratio Power 80 1 20 0.1 0.63 90% 80 1 20 0.3 0.78 59% 80 1 20 0.5 0.87 37% 60 1 40 0.1 0.40 >99.99% 60 1 40 0.3 0.62 91.4% 60 1 40 0.5 0.75 65.8%

Missing data. For those missing data the investigators will use intent-to-treat and multiple imputation (multiple imputation for chained equations [MICE]) using data on all observed baseline and outcome data.

Sample Size Re-Estimation. At the interim analysis (i.e., 50% of maximum enrollment), the investigators will estimate the CV, and re-estimate the required sample size. All analyses will either adjust for clinical site (e.g., in a regression model) or consider it as a stratification variable (e.g., in a Cochran-Mantel-Haenszel relative risk analysis).

SAS statistical software (Carey, North Carolina), R programming language (The R Project for Statistical Computing) and East 5.3 software (Cytel Inc.) will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of at least 18 years of age
2. A total of 1-6 traumatic rib fractures confirmed by imaging at least 3 cm distal to the costotransverse joint sustained within the previous 60 h (bilateral fractures are acceptable, but the total of the two sides combined must not exceed 6 fractures)
3. Pain in the fractured rib(s) region rated at least moderate (5 on the 0-10 Numeric Rating Scale) at rest
4. Undergoing a single-injection peripheral nerve block to treat the pain of the rib fracture(s)

Exclusion Criteria:

1. Anticoagulation or bleeding disorder: introduction of the percutaneous cryoneurolysis probe has a risk of hemorrhage similar to the percutaneous insertion of a similar gauge needle; but an anticoagulated state will increase the risk of hemorrhage (aspirin in doses for cardiothoracic/stroke prophylaxis [≤ 325 mg] are acceptable).
2. Infection at the site of probe introduction: percutaneous insertion of the probe through a cutaneous infection would bring an unacceptable risk of introducing the infection to deeper tissues.
3. Pulmonary disease or injury requiring supplemental oxygen: one theoretical risk of cryoneurolysis is a unilateral pneumothorax (not reported) which could result in a compromised pulmonary state for patients who require supplemental oxygen at baseline.
4. Neurologic deficit of the intercostal nerves of the fractured ribs: cryoneurolysis is theoretically a potent analgesic, but it does not "heal" injured nerves. Therefore, nerve deficits-either pre-existing or due to the trauma-will confound the analgesia-related results.
5. Possessing any contraindication to decreased temperature such as cryoglobulinemia, cryofibrinogenemia, cold urticaria paroxysmal cold hemoglobinuria, or Raynaud's disease: the decreased temperature accompanying cryoneurolysis could result in local tissue/vascular compromise for patients with any of these cold-triggered syndromes/diseases.
6. Insulin-dependent diabetes: laboratory studies have demonstrated impaired nerve regeneration in diabetic animals, and diabetes in patients can lead to impaired regeneration of axons and recovery following investigational nerve injury as well as focal neuropathies such as ulnar neuropathy and carpal tunnel syndrome. Whether these findings are applicable to cryoneurolysis in patients with diabetes remains unknown, but we prefer to error on the side of caution for study participants.
7. Chronic opioid use (daily use within the 2 weeks prior to the fracture and duration of use > 4 weeks): individuals using opioids on a chronic basis will continue their baseline opioid requirements following the traumatic event. This will confound the analgesic results of the study.
8. Inability to use an incentive spirometer: One of the Specific Aims involves improving functioning by decreasing pain using cryoneurolysis, and this will be evaluated using an incentive spirometer. For this reason, patients who are intubated or for whom there is anticipation of intubation will be excluded.
9. Any injury outside of the fractured rib(s) which results in moderate pain (NRS > 3) and/or anticipated to require opioid analgesics: such injuries would confound the results for the intervention under investigation.
10. An existing or planned continuous neuraxial or peripheral nerve block.
11. Fracture of the 1st rib on either side
12. Flail chest (3 or more adjacent ribs, each fractured in more than one location to create a free-floating segment)
13. Chest tube
14. Any degree of decreased mental capacity as determined by the surgical service or investigators.
15. Inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access).
16. Pregnancy
17. Incarceration
18. Number and location of fractures would require more than 10 intercostal nerves to be treated with cryoneurolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption during first 2 post-intervention months | Post-intervention months 1 and 2, collected on days 1, 2, 3, 7, 14, 21, 30, 45 and 60; at each collection time point, opioid use for the previous 24 hours will be recorded
  Cumulative opioid dose measured in oral oxycodone equivalents following intervention for 9 specific 24-hour time points over the first 2 months following surgery. With 9 time points (post-intervention days 1, 2, 3, 7, 14, 21, 30, 45 and 60), this will encompass 216 hours in total of the first 2 post-intervention months. In order to claim that percutaneous cryoneurolysis is superior to usual and customary analgesia, at least one of Outcomes 1 and 2 must be superior while the other at least noninferior.
Average pain during first 2 post-intervention months | Post-intervention months 1 and 2, collected on days 1, 2, 3, 7, 14, 21, 30, 45 and 60; at each collection time point, the "average" pain score for the previous 24 hours will be recorded
  The area under the curve for the "average" daily pain scores over the first 2 post-intervention months. At 9 specific time points the "average" pain score following the intervention will be measured using the numeric rating scale. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10= worst imaginable pain. In order to claim that percutaneous cryoneurolysis is superior to usual and customary analgesia, at least one of Outcomes 1 and 2 must be superior while the other at least noninferior.

SECONDARY OUTCOMES:
Opioid consumption | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  Cumulative opioid dose of the previous 24 hours measured in oral oxycodone equivalents
Average pain | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The "average" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Worst/maximum pain | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The "worst" or "maximum" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Least/lowest/minimal pain | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The "least" or "lowest" or "minimal" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Current pain | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The current pain level at the time of the data collection measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Brief Pain Inventory, short form (interference subscale) | Collected on post-intervention days 3, 7, 14, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
First 2 months area under the curve of the Brief Pain Inventory, short form (interference subscale) | Collected on post-intervention days 3, 7, 14, 30, 45 and 60
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale; (2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale. The secondary outcome of greatest interest will be the area under the curve for the interference domain collected over the first two months.
Pain during spirometry | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The pain level experienced while using the incentive spirometer measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Maximum voluntary inspiratory volume individual time points | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  We will follow the clinical guidelines published by the American Association for Respiratory Care: the spirometer is held in an upright position, the patient exhales completely, places the lips around the mouthpiece, inhales to the maximum volume over the course of 5 seconds, releases the mouthpiece and breath-holds, and then slowly exhales. This is repeated for a total of three times, and we will record the maximum volume for study purposes.
First 2 months area under the curve of the maximum voluntary inspiratory volume | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, 45, and 60
  We will follow the clinical guidelines published by the American Association for Respiratory Care: the spirometer is held in an upright position, the patient exhales completely, places the lips around the mouthpiece, inhales to the maximum volume over the course of 5 seconds, releases the mouthpiece and breath-holds, and then slowly exhales. This is repeated for a total of three times, and we will record the maximum volume for study purposes.
Awakenings due to pain | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  The number of times the patient awoke the previous night due to pain
Post-Traumatic Stress Disorder checklist (PCL-5) | Day of intervention (prior to intervention)
  A 20-item self-report measure reflecting symptoms of post-traumatic disorder validated in military, veteran and civilian populations.
Masking assessment | Post-intervention Day 7
  Whether or not the patient thinks they received the active cryoneurolysis recorded as "no", "yes", or "unsure"
Depression screening with the Patient Health Questionnaire (PHQ-2) | Post-intervention Months 3, 6, 9, and 12
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past 2 weeks, scoring each as 0 ("not at all") to 3 ("nearly every day"). The total score therefore ranges from 0-6 with a score of 3 most often used as a cut point when using the PHQ-2 to screen for major depression.
Nociceptive vs neuropathic pain estimation | Collected on post-intervention months 6, 9 and 12
  In patients who have a "worst" NRS>0 between 6-12 months, we will administer the self-report Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS). A score of 12 or more suggests pain of predominantly neuropathic origin.
Days hospitalized | Post-intervention Days 0-14
  Number of days from the intervention until the day of discharge measured in 1-day increments
Number of participants with pulmonary complications | Collected on post-intervention days 1, 2, 3, 7, 14, 21, 30, and 45; as well as months 2, 3, 6, 9, and 12
  Pulmonary complications will be recorded such as pneumonia, pneumothorax, hemothorax, pulmonary embolus, aspiration, empyema, acute respiratory distress syndrome, and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (5):
- United States (5):
  - University of California, San Diego, La Jolla, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Texas, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finneran Iv JJ, Gabriel RA, Swisher MW, Berndtson AE, Godat LN, Costantini TW, Ilfeld BM. Ultrasound-guided percutaneous intercostal nerve cryoneurolysis for analgesia following traumatic rib fracture -a case series. Korean J Anesthesiol. 2020 Oct;73(5):455-459. doi: 10.4097/kja.19395. Epub 2019 Nov 5. PMID 31684715
- [Background] Ilfeld BM, Finneran JJ. Cryoneurolysis and Percutaneous Peripheral Nerve Stimulation to Treat Acute Pain. Anesthesiology. 2020 Nov 1;133(5):1127-1149. doi: 10.1097/ALN.0000000000003532. PMID 32898231